CLINICAL TRIAL: NCT05159986
Title: Eefficacy of Diadynamic Currents Associated Exercise in Patients With Knee Osteoarthritis
Brief Title: Diadynamic and Exercises in Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CT01306435
Record Dates: First submitted 2021-11-10; First posted 2021-12-16 (Actual); Last update posted 2021-12-16 (Actual); Status verified 2021-11

CONDITIONS: Osteoarthritis, Knee
Keywords: PAIN; Electric Stimulation Therapy; Exercise Therapy
MeSH Terms: conditions — Osteoarthritis, Knee; Pain

STUDY DESIGN:
Intervention Model Description: Participants were randomly allocated to a Group I (diadynamic currents associated to Exercise; n=30, 60 knees) and Group II (exercises group; n=30, 60 knees) were treated 3 times a week for 8 weeks.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Diadynamic and Exercises (Experimental): Group Diadynamic and Exercises received Diadynamic currents associated to Exercise three times a week for 8 weeks following initial assessment (n=30, 60 knees) Diadynamic currents was performed with the following parameters: application of the two-phase current and then the long-term one. Each current was applied for 4 minutes on the medial and lateral sides of the knee.
  Interventions: Procedure: Group that received aplication of Diadynamic currents associated to Exercise during eight weeks with three sessions a week; Other: Group that received exercise during eight weeks with three sessions a week
- Group Exercises (Experimental): Group Exercises received only exercises three times a week for 8 weeks following initial assessment (n=30, 60 knees).
  Interventions: Other: Group that received exercise during eight weeks with three sessions a week

INTERVENTIONS:
Procedure: Group that received aplication of Diadynamic currents associated to Exercise during eight weeks with three sessions a week — Diadynamic currents was performed followed by exercises (divided into Phase-1, Phase-2 and Phase-3 during eight weeks with three sessions a week).
  Arms: Group Diadynamic and Exercises
Other: Group that received exercise during eight weeks with three sessions a week — The intervention was divided into Phase-1, Phase-2 and Phase-3 during eight weeks with three sessions a week. Each session lasted 45 minutes.

SUMMARY:
Osteoarthritis represents failed repair of joint damage resulting from stresses initiated by any joint or periarticular tissue abnormality. The rate of progression varies among persons and within a knee over time.

The symptoms and signs of knee osteoarthritis include pain, stiffness, reduced joint motion, and muscle weakness. Long-term consequences can include reduced physical activity, deconditioning, impaired sleep, fatigue, depression, and disability.This reduction in activity to avoid pain (kinesiophobia) to evade the onset of pain, especially in the acute phase, limiting their compliance with effective rehabilitation strategies such as regular exercises.

Physical medicine has a wide range of analgesic anti-inflammatory and muscle stimulating treatment methods. Both diadynamic and TENS currents have become the most frequently implemented electrotherapeutic methods. The impact of diadynamic currents consists of analgesic effects and specific dynamics during the formation of physiological processes in tissues.

They occur during the administration of the current and lasts up to a few hours after the treatment has been terminated. One of the theories explaining the analgesic effect of diadynamic currents is the gate control theory of pain by Wall and Melzack. Recently, another theory has become very popular. It explains the analgesic effect provoked by bodies characterized as polypeptides called endorphins. Electric stimulation using diadynamic currents generates an increase in the amount of endorphins in a system.

Although the analgesic impact of TENS therapy is well known, Diadynamic currents therapies have not been studied in knee osteoarthritis pain conditions. Therefore, the aim of the present study was to investigate the medium-term effects of Diadynamic currents combined with exercise on pain and disability in patients with osteoarthritis of the knee.

DETAILED DESCRIPTION:
The study included patients who attended the Special Rehabilitation Services in Taboão da Serra-SP, with knee osteoarthritis diagnosed by an independent rehabilitation specialist, and fulfilled the following inclusion criteria: (1) aged from 50 and 75; (2) symptomatic knee osteoarthritis for at least three months; (3) visual analogue scale12 score above 3 and (4) radiographic knee osteoarthritis (uni or bilateral) compatible with Kellgren-Lawrence grade two or higher.

The exclusion criteria were as follows: contraindication to laser application (e.g. cancer and insulin-dependent diabetes); inability to perform the assessment or treatment; continuous use of anti-inflammatory drugs, symptomatic hip osteoarthritis and physiotherapeutic knee treatment within the last 3 months.

All potentially eligible participants were contacted by telephone and those interested in participating were invited to attend a physical examination for inclusion and exclusion criterion. All participants were informed about the study and provided informed consent before participating. They were assigned by block randomization, stratified according to treatment group. An independent researcher not involved in outcome assessment was responsible for group allocation, using a computer-generated random number table. Immediately after baseline assessment by the blinded assessor, the treating physiotherapist accessed the allocation schedule from a centrally located locked cabinet. Patients and the physiotherapist responsible for the evaluation and physiotherapist responsible for the treatment were all unaware of the randomization results as allocation to groups was concealed.

Demographic and anthropometric data, the use of pain relief medications, the duration of knee pain, the knee range of motion, and a range of patient-reported outcomes were collected at baseline (before randomization) and 8 weeks from baseline by the same blinded evaluator.

The primary outcomes were pain intensity measured by the numeric pain rating scale (0-10) with a minimal clinically important change set at two points and disability measured using the Lequesne questionnaire, which consists of 11 questions about pain, discomfort, and function. Scores range from 0 to 24 (from 'no' to 'extremely severe' dysfunction).

Secondary outcomes included medication intake (Paracetamol) for knee pain relief, mobility and balance, range of motion, muscular strength, and activity. Mobility and balance were evaluated by the Timed Up and Go test. The Timed Up and Go test, a measure of functional mobility, quantifies in seconds the time that the individual needs to stand up from a chair, walk 3m, turn back toward the chair and sit down again. Range of motion of the knees was measured with a universal goniometer (AESCULAP). Muscular strength was estimated at maximal isometric force for the quadriceps, using a portable dynamometer (Lafayette, USA). Under stabilized conditions, patients, sitting with knees flexed at 60 (measured by a goniometer), were asked to extend the legs as far as they could. Three attempts were conducted, and the mean value was obtained. Muscular strength was estimated at maximal isometric force for the quadriceps, using a portable dynamometer. Under stabilized conditions, patients, sitting with knees flexed at 10, 60 and 90 degrees (measured by a goniometer), were asked to extend the legs as far as they could. Three attempts were conducted and the mean value was obtained. Physical activity was measured using the Western Ontario and McMaster Universities Osteoarthritis questionnaire, which is self-administered and measures pain, stiff joints, and physical activity. Increased scores suggest decreased activity.

In this study, all patients had osteoarthritis of both knees, and in every patient both knees were treated with the allocated treatment.

Participants in the Group I received Diadynamic currents associated to Exercise while the Group II received only exercises three times a week for 8 weeks following initial assessment.

The group I, Diadynamic currents was performed with the following parameters: application of the two-phase current and then the long-term one. Each current was applied for 4 minutes on the medial and lateral sides of the knee.

All patients followed the same training program (Table 1). The intervention was divided into Phase-1, Phase-2 and Phase-3 during eight weeks with three sessions a week. Each session lasted 45 minutes:

* 10 minutes warming-up (treadmill, ergometer bike or rowing machine);
* 30 minutes 2-3 sets with Phase-1, Phase-2 and Phase-3;
* 5 minutes stretching (hamstrings, quadriceps, adductors, and gastrocmenius). Participants were instructed not to use analgesic medications other than paracetamol (500 mg/day) or anti-inflammatory drugs during the study, and not to perform any other type of physical exercise in addition to the exercise performed during the study.

After describing the data, the hypothesis of normality of continuous variables was tested using the Shapiro-Wilk test. The age, weight, height and BMI of volunteers between groups were compared using Student's t-test for independent samples. To investigate the effect of the treatment on the pre and post evaluation, as well as the interaction of this effect between the groups, the General Linear Models with mixed design (evaluations x groups) were applied. To analyze the effects of the interactions, Tukey's Post Hoc tests were performed considering an alpha error of 5%. All analyzes were performed using the statistical program R version 3.1.3 using the R Commander graphical interface.

ELIGIBILITY:
Inclusion Criteria:

1. aged from 50 and 75;
2. symptomatic knee osteoarthritis for at least three months;
3. visual analogue scale12 score above 3 and
4. radiographic knee osteoarthritis (uni or bilateral) compatible with Kellgren-Lawrence13 grade two or higher.

Exclusion Criteria:

1. contraindication to laser application (e.g. cancer and insulin-dependent diabetes);
2. inability to perform the assessment or treatment;
3. continuous use of anti-inflammatory drugs,
4. symptomatic hip osteoarthritis
5. physiotherapeutic knee treatment within the last 3 months.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Change in pain intensity | outcomes were collected at baseline (before randomization) and 8 weeks from baseline by the same blinded evaluator.
  Pain intensity measured by the numeric pain rating scale (0-10) with a minimal clinically important change set at two points
Change in Disability | outcomes were collected at baseline (before randomization) and 8 weeks from baseline by the same blinded evaluator.
  Disability measured using the Lequesne questionnaire,14 which consists of 11 questions about pain, discomfort, and function. Scores range from 0 to 24 (from 'no' to 'extremely severe' dysfunction).

SECONDARY OUTCOMES:
Change in Medication intake (Paracetamol) for knee pain relief | outcomes were collected at baseline (before randomization) and 8 weeks from baseline by the same blinded evaluator.
  Control of the use of pain medications before, during and after treatment.
Change in Mobility and balance | outcomes were collected at baseline (before randomization) and 8 weeks from baseline by the same blinded evaluator.
  Mobility and balance were evaluated by the Timed Up and Go test. The Timed Up and Go test, a measure of functional mobility, quantifies in seconds the time that the individual needs to stand up from a chair, walk 3m, turn back toward the chair and sit down again.
Change in Range of motion | outcomes were collected at baseline (before randomization) and 8 weeks from baseline by the same blinded evaluator.
  Range of motion of the knees was measured with a universal goniometer (AESCULAP).
Change in Muscular strength | outcomes were collected at baseline (before randomization) and 8 weeks from baseline by the same blinded evaluator.
  Muscular strength was estimated at maximal isometric force for the quadriceps, using a portable dynamometer (Lafayette, USA). Under stabilized conditions, patients, sitting with knees flexed at 60 (measured by a goniometer),17 were asked to extend the legs as far as they could. Three attempts were conducted, and the mean value was obtained. Muscular strength was estimated at maximal isometric force for the quadriceps, using a portable dynamometer. Under stabilized conditions, patients, sitting with knees flexed at 10, 60 and 90 degrees (measured by a goniometer),17 were asked to extend the legs as far as they could. Three attempts were conducted and the mean value was obtained.
Change in Physical activity | outcomes were collected at baseline (before randomization) and 8 weeks from baseline by the same blinded evaluator.
  Physical activity was measured using the Western Ontario and McMaster Universities Osteoarthritis questionnaire,18 which is self-administered and measures pain, stiff joints, and physical activity. Increased scores suggest decreased activity.

CONTACTS AND LOCATIONS:
Overall Officials: Raquel Ap Casarotto, PhD, Principal Investigator — USP
Locations (1):
- Raquel Aparecida Casarotto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No